CLINICAL TRIAL: NCT00953121
Title: Phase II Study of Bevacizumab Plus Irinotecan and Carboplatin for Recurrent Malignant Glioma Patients
Brief Title: Bevacizumab Plus Irinotecan Plus Carboplatin for Recurrent Malignant Glioma (MG)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Annick Desjardins (Other)
Responsible Party: Sponsor-Investigator, Annick Desjardins, Assist Professor of Medicine-Neurology, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00016712
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Results first posted 2013-09-04 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2013-09

CONDITIONS: Malignant Glioma
Keywords: irinotecan; carboplatin; bevacizumab; Avastin
MeSH Terms: conditions — Glioma | interventions — Bevacizumab; Irinotecan; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort A-Grade IV No Failure (Experimental): Recurrent GBM patients who have not previously failed bevacizumab, irinotecan, or carboplatin
  Interventions: Drug: bevacizumab and CPT-11 and Carboplatin
- Cohort B-Grade III No Failure (Experimental): Recurrent Grade 3 malignant glioma patients who have not previously failed either bevacizumab, irinotecan or carboplatin
  Interventions: Drug: bevacizumab and CPT-11 and Carboplatin
- Cohort C-Failed Prior Therapy (Experimental): Recurrent Grade IV GBM patients who have failed prior bevacizumab therapy, but not prior CPT-11 or carboplatin therapies
  Interventions: Drug: bevacizumab and CPT-11 and Carboplatin

INTERVENTIONS:
Drug: bevacizumab and CPT-11 and Carboplatin — Bevacizumab will be administered at 10mg/kg with irinotecan every other week. The dose of irinotecan will be 125 mg/m2 for patients not on CYP3A-inducing anti=epileptics (EIAEDs) and 340 mg/m2 for patients on EIAEDs. All patients will also receive carboplatin on day 1 of each 28-day treatment cycle. Carboplatin will be dosed to achieve an AUC of 4.
  Other Names: bevacizumab; Avastin; Irinotecan; CPT-11; Carboplatin; Paraplatin; Camptosar

SUMMARY:
The purpose of this study is to determine whether Bevacizumab, CPT-11 and Carboplatin in combination are effective in the treatment of recurrent malignant glioma.

DETAILED DESCRIPTION:
Three cohorts will accrue and will be assessed independently. Each cohort will evaluate a separate malignant glioma subpopulation. Cohort A will assess recurrent glioblastoma multiforme (GBM) subjects who have not previously failed either bevacizumab, irinotecan or carboplatin. Cohort B will assess recurrent grade 3 malignant glioma subjects who have not previously failed either bevacizumab, irinotecan or carboplatin. Cohort C will assess recurrent GBM subjects who have failed prior bevacizumab therapy but who have not failed prior irinotecan or carboplatin. The primary endpoint of each cohort will be 6-month progression-free survival. This study will be conducted at The Preston Robert Tisch Brain Tumor Center at Duke.

For each cohort, bevacizumab will be administered at 10 mg/kg with irinotecan every other week. The dose of irinotecan will be 125 mg/m2 for subjects not on Cytochrome P450, family 3, subfamily A (CYP3A)-inducing anti-epileptics (EIAEDs) and 340 mg/m2 for subjects on EIAEDs. All subjects will also receive carboplatin on day 1 of each 28-day treatment cycle. Carboplatin will be dosed to achieve an area under the curve (AUC) of 4.

Within 2 weeks of starting the study, subject's medical history and current medical conditions will be recorded. A physical examination including vital signs (temperature, respiratory rate, blood pressure, and pulse), height and weight, and neurological examination will be done. Subject will be asked about his or her ability to perform everyday tasks. Blood tests for assessment of a complete blood count including monitoring liver and kidney function and a urine test to check kidney function will be performed. For women of childbearing potential, a blood test to rule out pregnancy will be done prior to the start of treatment. Blood tests will also check for a specific gene, which may affect how much irinotecan subject is given. A magnetic resonance imaging (MRI) of will be performed within 2 weeks before starting study drugs as well as after every eight weeks to determine response and progression.

In total, approximately 3 teaspoons (15 mL) of blood will be drawn for the evaluations before starting study drug. These tests will be repeated every 8 weeks (blood chemistries), except a complete blood count (approximately 1 teaspoon), which will need to be repeated every week as well as when it is deemed clinically necessary to repeat. Every 4 weeks a urine test will be performed to test the amount of protein in subject's urine.

Placement of a central venous line may be required. Subjects will be seen in the clinic for a physical and neurological examination every four (4) weeks. Urine and blood laboratory tests will also be obtained at these visits. In addition, a complete blood count (about 1 teaspoon) will be obtained every week. Blood pressure measurement will be required every 2 weeks. MRI (Magnetic Resonance Imaging) scans will be done every 8 weeks (after every 2 cycles) to determine the effectiveness of the study drugs. If the tumor remains the same size or smaller, subject will continue to receive study drugs for 12 cycles unless there are bad side effects or unless there is evidence that the drug is not working. If evaluations show that there may be persistent tumor after 12 cycles, subject may continue treatment. Study drugs will stop if the subject's tumor gets larger.

Additional tests may be done at the discretion of the doctor as part of regular care throughout the study. These exams and tests will be done to monitor the effects of the study interventions.

ELIGIBILITY:
Inclusion Criteria:

Cohorts A and B only

* No prior failure or grade ≥ 3 toxicity to bevacizumab, irinotecan or carboplatin.

Cohort C only

* Failure on prior bevacizumab therapy
* No prior failure or grade ≥ 3 toxicity to either irinotecan or carboplatin.

All Cohorts

* Age * 18 years
* Karnofsky Performance Status (KPS) ≥ 70%
* No more than 3 prior episodes of disease progression
* An interval of at least 4 weeks between prior surgical resection or one week from stereotactic biopsy
* An interval of at least 12 weeks from the end of prior radiotherapy unless there is a new area of enhancement consistent with recurrent tumor outside of the radiation field, or there are progressive changes on MRI on at least two consecutive MRI scans at least four weeks apart, or there is biopsy-proven tumor progression
* An interval of at least 4 weeks from prior chemotherapy (6 weeks for nitrosoureas) or investigational agent unless the patient has recovered from all anticipated toxicities associated with that therapy
* Hematocrit ≥ 29%, absolute neutrophil count (ANC) ≥ 1,000 cells/*l, platelets ≥ 100,000 cells/*l
* Serum creatinine ≤ 1.5 times upper limit of normal, serum glutamic oxaloacetic transaminase (SGOT) ≤ 2.5 times upper limit of normal and bilirubin ≤ 2.0 times upper limit of normal
* International Normalized Ratio (INR) < 1.5 or prothrombin time/partial thromboplastin time (PT/PTT) within 1.5 time upper limit of normal (ULN).
* Signed informed consent approved by the Institutional Review Board prior to patient entry
* No evidence of hemorrhage on the baseline MRI or CT scan other than those that are stable grade 1
* If sexually active, patients will take contraceptive measures for the duration of the treatments. Medically acceptable contraceptives include: (1) surgical sterilization (such as a tubal ligation, hysterectomy, vasectomy), (2) approved hormonal contraceptives (such as birth control pills, patches, implants or injections), (3) barrier methods (such as a condom or diaphragm) used with a spermicide, or (4) an intrauterine device (IUD)

Exclusion Criteria:

Disease-Specific Exclusions

* Co-medication that may interfere with study results; e.g. immuno-suppressive agents other than corticosteroids
* Active infection requiring intravenous antibiotics
* Requires therapeutic anti-coagulation with warfarin

General Medical Exclusions

Subjects meeting any of the following criteria are ineligible for study entry:

* Inability to comply with study and/or follow-up procedures
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored bevacizumab cancer study
* Severe hepatic insufficiency (ongoing grade 3 or greater hepatic adverse events) or known active chronic hepatitis
* Homozygosity for the *28 uridine diphosphate glucuronosyltransferase 1A1 (UGT1A1) allele.

Bevacizumab-Specific Exclusions

* Inadequately controlled hypertension (defined as systolic blood pressure > 150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications)
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 6 months prior to study enrollment
* History of stroke or transient ischemic attack within 6 months prior to study enrollment
* Significant vascular disease (e.g., aortic aneurysm, aortic dissection)
* Symptomatic peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
* Serious, non-healing wound, ulcer, or bone fracture
* Proteinuria at screening as demonstrated by either:
* Urine protein:creatinine (UPC) ratio ≥ 1.0 at screening OR
* Urine dipstick for proteinuria ≥ 2+ (patients discovered to have ≥2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible)
* Known hypersensitivity to any component of bevacizumab, Chinese hamster ovary cell products or other recombinant human or humanized antibodies."
* Pregnant (positive pregnancy test) or lactating. Use of effective means of contraception (men and women) in subjects of child-bearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2009-09; Primary Completion 2012-07 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annick Desjardins, MD, FRCPC, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

REFERENCES:
- [Derived] Reardon DA, Desjardins A, Peters KB, Gururangan S, Sampson JH, McLendon RE, Herndon JE 2nd, Bulusu A, Threatt S, Friedman AH, Vredenburgh JJ, Friedman HS. Phase II study of carboplatin, irinotecan, and bevacizumab for bevacizumab naive, recurrent glioblastoma. J Neurooncol. 2012 Mar;107(1):155-64. doi: 10.1007/s11060-011-0722-2. Epub 2011 Oct 11. PMID 21986722
- See also: The Preston Robert Tisch Brain Tumor Center at DUKE — http://www.cancer.duke.edu/btc/

RESULTS

PARTICIPANT FLOW:
Groups:
- Grade IV, No Bevacizumab Failure: Recurrent Glioblastoma Multiforme (GBM) patients who have not previously failed bevacizumab, irinotecan, or carboplatin
  bevacizumab and CPT-11 and Carboplatin : Bevacizumab will be administered at 10mg/kg with irinotecan every other week. The dose of irinotecan will be 125 mg/m2 for patients not on CYP3A-inducing anti=epileptics (EIAEDs) and 340 mg/m2 for patients on EIAEDs. All patients will also receive carboplatin on day 1 of each 28-day treatment cycle. Carboplatin will be dosed to achieve an area under the curve (AUC) of 4.
- Grade III, No Bevacizumab Failure: Recurrent Grade 3 malignant glioma patients who have not previously failed either bevacizumab, irinotecan or carboplatin
  bevacizumab and CPT-11 and Carboplatin : Bevacizumab will be administered at 10mg/kg with irinotecan every other week. The dose of irinotecan will be 125 mg/m2 for patients not on CYP3A-inducing anti=epileptics (EIAEDs) and 340 mg/m2 for patients on EIAEDs. All patients will also receive carboplatin on day 1 of each 28-day treatment cycle. Carboplatin will be dosed to achieve an AUC of 4.
- Grade IV, Bevacizumab Failure: Recurrent Grade IV GBM patients who have failed prior bevacizumab therapy, but not prior CPT-11 or carboplatin therapies
  bevacizumab and CPT-11 and Carboplatin : Bevacizumab will be administered at 10mg/kg with irinotecan every other week. The dose of irinotecan will be 125 mg/m2 for patients not on CYP3A-inducing anti=epileptics (EIAEDs) and 340 mg/m2 for patients on EIAEDs. All patients will also receive carboplatin on day 1 of each 28-day treatment cycle. Carboplatin will be dosed to achieve an AUC of 4.
Period: Overall Study
Arm/Group | Grade IV, No Bevacizumab Failure | Grade III, No Bevacizumab Failure | Grade IV, Bevacizumab Failure
Started | 40 | 39 | 25
Completed | 40 | 39 | 25
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Grade IV, No Bevacizumab Failure: Recurrent GBM patients who have not previously failed bevacizumab, irinotecan, or carboplatin
  bevacizumab and CPT-11 and Carboplatin : Bevacizumab will be administered at 10mg/kg with irinotecan every other week. The dose of irinotecan will be 125 mg/m2 for patients not on CYP3A-inducing anti=epileptics (EIAEDs) and 340 mg/m2 for patients on EIAEDs. All patients will also receive carboplatin on day 1 of each 28-day treatment cycle. Carboplatin will be dosed to achieve an AUC of 4.
- Total: Total of all reporting groups
Arm/Group | Grade IV, No Bevacizumab Failure | Grade III, No Bevacizumab Failure | Grade IV, Bevacizumab Failure | Total
Number analyzed (Participants) | 40 | 39 | 25 | 104
Age Continuous [Median (Full Range); unit: years] | 51 [25 to 72] | 47 [26 to 71] | 52 [19 to 76] | 50 [19 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 8 | 29
  Male | 30 | 28 | 17 | 75

OUTCOME MEASURES:

1. Primary Outcome: 6 Month Progression-free Survival
Description: Percentage of participants surviving six months from the start of study treatment without progression of disease. PFS was defined as the time from the date of study treatment initiation to the date of the first documented progression according to the Response Assessment in Neuro-Oncology (RANO) criteria, or to death due to any cause. Progression is defined as greater than or equal to a 25% increase in the product of the largest perpendicular diameters of any enhancing lesion or any new enhancing tumor on MRI scans. Patients may also be classified as progressive disease with significant neurologic decline felt to be due to underlying tumor and not attributable to co-morbid event or concurrent medication regardless of MRI findings.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Grade IV, No Bevacizumab Failure | Grade III, No Bevacizumab Failure | Grade IV, Bevacizumab Failure
Number analyzed (Participants) | 40 | 39 | 25
percentage of participants | 47.5 [31.6 to 61.8] | 71.1 [53.9 to 82.8] | 24.0 [9.8 to 41.7]

2. Secondary Outcome: Objective Response Rate
Description: Percentage of participants with an objective response (complete response or partial response) based on Response Assessment in Neuro-Oncology (RANO) criteria. A complete response is defined as disappearance of all enhancing tumor on contrast enhanced MRI scan. Patient must be off steroids or only on adrenal maintenance doses. A partial response is defined as greater than or equal to a 50% reduction in the size (products of the largest perpendicular diameters) for all enhancing lesions. No new lesions may arise. Steroids must be stable or decreasing dose.
Time Frame: 34 months
Population: The number of participants analyzed is lower than the total number in the study for each arm due to the fact that some patients progressed or experienced an adverse event which resulted in being taken off study during the first cycle and thus were never evaluated for radiographic response.
Measure: Number; unit: participants
Arm/Group | Grade IV, No Bevacizumab Failure | Grade III, No Bevacizumab Failure | Grade IV, Bevacizumab Failure
Number analyzed (Participants) | 35 | 36 | 24
participants | 0 | 0 | 0

3. Secondary Outcome: Median Progression Free Survival (PFS)
Description: Time in months from the start of study treatment to the date of first progression according to RANO criteria, or to death due to any cause. Patients alive who had not progressed as of the last follow-up had PFS censored at the last follow-up date. Median PFS was estimated using a Kaplan-Meier curve.
Time Frame: 40 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Grade IV, No Bevacizumab Failure | Grade III, No Bevacizumab Failure | Grade IV, Bevacizumab Failure
Number analyzed (Participants) | 40 | 39 | 25
months | 5.9 [4.8 to 8.5] | 10.0 [7.3 to 12.1] | 3.6 [2.7 to 4.3]

4. Secondary Outcome: Median Overall Survival (OS)
Description: Time in months from the start of study treatment to date of death due to any cause. Patients alive as of the last follow-up had OS censored at the last follow-up date. Median OS was estimated using a Kaplan-Meier curve.
Time Frame: 40 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Grade IV, No Bevacizumab Failure | Grade III, No Bevacizumab Failure | Grade IV, Bevacizumab Failure
Number analyzed (Participants) | 40 | 39 | 25
months | 9.3 [7.0 to 11.9] | 16.0 [12.2 to 21.9] | 5.9 [4.0 to 8.5]

5. Secondary Outcome: Safety of Bevacizumab (Avastin) in Combination With Irinotecan and Carboplatin
Description: Number of patients experiencing a toxicity greater than or equal to grade 2 treatment-related toxicity
Time Frame: 34 months
Measure: Number; unit: participants
Arm/Group | Grade IV, No Bevacizumab Failure | Grade III, No Bevacizumab Failure | Grade IV, Bevacizumab Failure
Number analyzed (Participants) | 40 | 39 | 25
participants | 39 | 39 | 23

ADVERSE EVENTS:
Time Frame: 34 months
Description: The adverse events were gathered in Common Terminology Criteria for Adverse Events v.3.0, and have been converted to v.4.0 for entry into ClinicalTrials.gov
Arm/Group | Grade IV, No Bevacizumab Failure | Grade III, No Bevacizumab Failure | Grade IV, Bevacizumab Failure
Serious Adverse Events (participants affected / at risk) | 17/40 | 10/39 | 6/25
Other Adverse Events (participants affected / at risk) | 34/40 | 37/39 | 21/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Grade IV, No Bevacizumab Failure (N=40) | Grade III, No Bevacizumab Failure (N=39) | Grade IV, Bevacizumab Failure (N=25)
Anemia (Blood and lymphatic system disorders) | 2 | 1 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Colonic perforation (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal disorders - Other, specify: Fistula, GI: Small bowel NOS (Gastrointestinal disorders) | 1 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Death NOS (General disorders) | 7 | 1 | 0
Fatigue (General disorders) | 1 | 1 | 1
Sudden death NOS (General disorders) | 0 | 1 | 0
Esophageal infection (Infections and infestations) | 1 | 0 | 0
Infections and infestations - Other, specify: Infection with Gr 3 or 4 neutrophils: Lung (pneumonia) (Infections and infestations) | 1 | 0 | 0
Infections and infestations - Other, specify: Infection with Gr 3 or 4 neutrophils: Pharynx (Infections and infestations) | 0 | 1 | 0
Infections and infestations - Other, specify: Infection with Gr 3, 4 neutrophils: Skin (cellulitis) (Infections and infestations) | 0 | 0 | 1
Infections and infestations - Other, specify: Infection with Gr 3 or 4 neutrophils: Trachea (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 1 | 0
Meningitis (Infections and infestations) | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 1 | 0
Creatinine increased (Investigations) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 2 | 2 | 0
Platelet count decreased (Investigations) | 2 | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 0 | 1
Cognitive disturbance (Nervous system disorders) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Intracranial hemorrhage (Nervous system disorders) | 1 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 2 | 0 | 0
Seizure (Nervous system disorders) | 4 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1
Thromboembolic event (Vascular disorders) | 1 | 3 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Grade IV, No Bevacizumab Failure (N=40) | Grade III, No Bevacizumab Failure (N=39) | Grade IV, Bevacizumab Failure (N=25)
Anemia (Blood and lymphatic system disorders) | 8 | 7 | 4
Palpitations (Cardiac disorders) | 0 | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 0
Optic nerve disorder (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 7 | 2
Diarrhea (Gastrointestinal disorders) | 7 | 6 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal disorders - Other, specify: Gastroesophageal Reflux (Gastrointestinal disorders) | 1 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 2 | 0
Mucositis oral (Gastrointestinal disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 7 | 15 | 6
Oral hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 5 | 3
Edema limbs (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 21 | 23 | 6
Injection site reaction (General disorders) | 0 | 2 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Immune system disorders - Other, specify: Infusion reaction to CPT-11 (Immune system disorders) | 0 | 1 | 0
Bronchial infection (Infections and infestations) | 1 | 0 | 0
Infections and infestations - Other, specify: Infection with normal ANC - Herpes Zoster (Infections and infestations) | 0 | 1 | 0
Infections and infestations - Other, specify: Shingles (Infections and infestations) | 1 | 0 | 0
Joint infection (Infections and infestations) | 1 | 0 | 0
Lip infection (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0
Upper respiratory infection (Infections and infestations) | 5 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 3 | 2 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 1
Neutrophil count decreased (Investigations) | 22 | 24 | 19
Platelet count decreased (Investigations) | 13 | 17 | 12
Weight loss (Investigations) | 0 | 0 | 2
White blood cell decreased (Investigations) | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 5 | 3 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 3 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | 6 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specify: Leg cramping during infusions (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 2
Dysphasia (Nervous system disorders) | 1 | 2 | 1
Headache (Nervous system disorders) | 8 | 5 | 1
Intracranial hemorrhage (Nervous system disorders) | 1 | 1 | 0
Ischemia cerebrovascular (Nervous system disorders) | 0 | 3 | 0
Nervous system disorders - Other, specify: Infusion Reaction (Nervous system disorders) | 0 | 1 | 0
Nervous system disorders - Other, specify: Neuropathy - Peripheral (Nervous system disorders) | 0 | 1 | 0
Nervous system disorders - Other, specify: Reaction to Carboplatin (Nervous system disorders) | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 7 | 11 | 4
Syncope (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 0
Confusion (Psychiatric disorders) | 0 | 1 | 1
Depression (Psychiatric disorders) | 3 | 4 | 1
Insomnia (Psychiatric disorders) | 2 | 0 | 0
Proteinuria (Renal and urinary disorders) | 3 | 2 | 4
Renal and urinary disorders - Other, specify: Kidney Stones (causing 3+ hematuria) (Renal and urinary disorders) | 0 | 1 | 0
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Hot flashes (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 2 | 3 | 2
Hypotension (Vascular disorders) | 0 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 2 | 0
Thromboembolic event (Vascular disorders) | 1 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes